CLINICAL TRIAL: NCT01302977
Title: Tracheal Occlusion Guided by Percutaneous Fetoscopy in Fetuses With Severe Isolated Congenital Diaphragmatic Hernia
Brief Title: Fetal Tracheal Occlusion in Severe Diaphragmatic Hernia: a Randomized Trial
Acronym: BRAFETO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Rodrigo Ruano, MD, PhD, Faculdade de Medicina da Universidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPPesq 1087/07
Record Dates: First submitted 2011-02-21; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Congenital Diaphragmatic Hernia; Congenital Abnormality
Keywords: Congenital diaphragmatic hernia; Fetal anomalies
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Congenital Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fetal intervention (Experimental): Composed of fetuses that undergo to fetal tracheal occlusion at 26-28 weeks.
  Interventions: Procedure: Fetal tracheal occlusion
- Control (No Intervention): Composed of fetuses that do not undergo fetal intervention

INTERVENTIONS:
Procedure: Fetal tracheal occlusion — Insertion of a detachable balloon inside fetal trachea by percutaneous fetoscopy
  Other Names: FETO, TO
  Arms: Fetal intervention

SUMMARY:
The neonatal mortality rate in cases with severe isolated congenital diaphragmatic hernia is higher than 90% due to severe pulmonary hypoplasia. Many studies have suggested that fetal tracheal occlusion may increase lung volumes and therefore reducing the risk for severe pulmonary hypoplasia and by consequence the risk for neonatal death.

The main objective of the present study is to evaluate if fetal tracheal occlusion improves survival rate in those cases that are followed in our hospital, by conducing a randomized trial.

DETAILED DESCRIPTION:
Fetuses will be randomly allocated in two groups: 1. for fetal tracheal occlusion at 26-28 weeks (FETO group) or 2. Postnatal therapy only (Control)

Main outcome: Survival rate in both groups Second outcomes: Postnatal diagnosis of severe pulmonary arterial hypertension, percentage of newborns in each group that will have clinical conditions for neonatal surgical repair of the diaphragmatic defect, fetal lung responses (increase of fetal lung size), maternal and obstetrical complications (prematurity, preterm rupture of the membranes, maternal hemorrhage and infection).

ELIGIBILITY:
Inclusion Criteria:

* ultrasound diagnosis of congenital diaphragmatic hernia
* fetuses at gestational age between 24 and 28 weeks
* absence of chromosomal and/or other structural anomalies (isolated congenital diaphragmatic hernia)
* severe congenital diaphragmatic hernia defined by lung-head ratio < 1.0 and more than 1/3 of liver herniated into fetal thorax and observed/expected fetal total lung volume < 0.35
* patient's consent to participate in the present study

Exclusion Criteria:

* Patient's refusal to participate in the study after allocation
* Preterm labor diagnosed before the procedure
* Preterm rupture of membranes before fetal intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 year
  Noenatal survival rate which includes percentage of newborns that survive up to 30 days of life.
  Infant survival rate which includes percentage of newborns that survive up to one year of life. Outcome measurement will be assessed up to one year after birth.

SECONDARY OUTCOMES:
Postnatal pulmonary arterial hypertension | 30 days of life
  Postnatal pulmonary arterial hypertension will be assessed up to 30 days of life according to the echocardiographic findings.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, MD, PhD, Principal Investigator — Faculdade de Medicina da Universidade de Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ruano R, Duarte SA, Pimenta EJ, Takashi E, da Silva MM, Tannuri U, Zugaib M. Comparison between fetal endoscopic tracheal occlusion using a 1.0-mm fetoscope and prenatal expectant management in severe congenital diaphragmatic hernia. Fetal Diagn Ther. 2011;29(1):64-70. doi: 10.1159/000311944. Epub 2010 Apr 10. PMID 20389048
- [Derived] Ruano R, Yoshisaki CT, da Silva MM, Ceccon ME, Grasi MS, Tannuri U, Zugaib M. A randomized controlled trial of fetal endoscopic tracheal occlusion versus postnatal management of severe isolated congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2012 Jan;39(1):20-7. doi: 10.1002/uog.10142. Epub 2011 Dec 14. PMID 22170862